CLINICAL TRIAL: NCT00275717
Title: The Effects of Thymoglobulin on Antibody Screening Cells.
Brief Title: A Study That Will Look at the Impact of Immunosuppression on Antibody Production in Kidney Transplant Recipients.
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Mark D. Stegall, MD, Mayo Clinic
Other Study IDs: 374-05
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-12

CONDITIONS: Kidney Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study is being done to collect blood and bone marrow samples for biologic studies of antibody producing cells. Donor specific antibodies can cause damage to the kidneys after they are transplanted. The study will look at the impact of immunosuppression on antibody production by antibody producing cells.

DETAILED DESCRIPTION:
Bone marrow and blood samples from both non-sensitized kidney transplant recipients and sensitized kidney transplant recipients will be collected. The samples will be used to compare the effect immunosuppression has on the antibody producing cells from both of these kinds of transplant recipients. Bone marrow will be collected from sensitized kidney transplant recipients before desensitization therapy prior to transplantation and at the time of kidney transplant surgery. Non-sensitized patients will have bone marrow collected only at the time of kidney transplant surgery. Blood will be collected at the same time point that the marrow is collected in both kinds of patients.

ELIGIBILITY:
Participants must be between the ages of 18 and 70 years of age and undergoing a kidney transplant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three groups will be studied:
  1. Non-sensitized renal allograft candidates prior to any therapy;
  2. High DSA recipients--Recipients with a positive T or B cell cytotoxicity crossmatch or a B cell flow cytometric crossmatch assay with a channel shift >350 at baseline against their living donor at baseline and
  3. Low DSA recipients-recipients with a negative T and B cell cytotoxicity assay, but a positive T or B cell flow cytometric crossmatch with a B cell channel shift <350.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2005-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Stegall, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States